CLINICAL TRIAL: NCT06993480
Title: A Single-Center, Open-Label Phase II Clinical Study to Evaluate the Antiviral Activity and Immune Responses of AHB-137 Injection in Participants With CHB Treated With Nucleos (t) Ide Analogues
Brief Title: A Study to Evaluate the Antiviral Activity and Immune Response of AHB-137 Injection in Participants With Chronic Hepatitis B (CHB)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ausper Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-10-8005
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AHB-137 (Experimental): AHB-137 will be injected subcutaneously.
  Interventions: Drug: AHB-137

INTERVENTIONS:
Drug: AHB-137 — AHB-137 300 mg will be injected subcutaneously once a week (total 24 weeks).

SUMMARY:
AB-10-8005 is a single-center, open-label Phase II clinical study to evaluate the antiviral activity and immune responses of AHB-137 injection in participants with CHB treated with nucleos (t) ide analogues.

DETAILED DESCRIPTION:
The study is to evaluate the antiviral activity and immune response of AHB-137 injection in participants with CHB treated with nucleos(t)ide analogues. The study is proposed to enroll 20-30 patients, with a total study duration of approximately 56 weeks per participants, including a screening period (up to 4 weeks), a clinical study lead-in period (approximately 4 weeks), an AHB-137 treatment period (24 weeks) and a follow-up period (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participated in the study and signed an informed consent form;
* Aged between 18 and 55 years at the time of signing the informed consent form;
* Body mass index (BMI) within the range of 18-30 kg/ m2;
* HBeAg negative or positive at screening;
* HBsAg or HBV DNA positive for at least 6 months;
* Have been on continuous nucleos(t)ide analogues antiviral therapy for more than 6 months prior to screening;
* 100 IU/mL < HBsAg ≤ 3000 IU/mL and HBV DNA < 100 IU/mL at screening;
* Alanine aminotransferase (ALT) ≤ 2 × upper limit of normal (ULN);
* Effective contraception as required.

Exclusion Criteria:

* Clinically significant abnormalities other than a history of CHB infection;
* Concomitant clinically significant other liver diseases;
* Any serious infection other than CHB infection requiring intravenous anti-infective therapy within 1 month prior to screening;
* Active hepatitis C, Human immunodeficiency virus (HIV) positive, syphilis positive;
* Liver stiffness value (LSM) > 9.0 kPa at screening;
* Diagnosis or suspicion of hepatocellular carcinoma, or alpha-fetoprotein (AFP) concentration ≥ 20 ng/mL at screening;
* Participants with confirmed or suspected hepatic decompensated hepatitis B cirrhosis;
* Liver biopsy at screening assessed severity of activity ≥ G3 grade and/or fibrosis reaching S4 stage;
* History of extrahepatic disease possibly related to HBV immune status;
* Ongoing or taking any immunosuppressive medication within 3 months prior to screening. Those who have used immunomodulators and cytotoxic drugs within 6 months prior to the first dose, or have a history of vaccination within 1 month prior to screening or have a live vaccination plan during the trial; Continuous use of traditional Chinese medicine for more than 2 months within 1 year prior to screening, or within 1 month prior to screening; Ongoing use of anticoagulants, bleeding tendency or coagulopathy, or conditions that, in the opinion of the investigator, increase the risk of liver biopsy;
* Receiving or using any interferon-containing therapy within 12 months prior to screening;
* History of malignancy within 5 years prior to screening or being evaluated for possible malignancy;
* Suspected history of allergy to any component of the study drug, or allergic constitution (multiple drug and food allergy, and judged by the investigator to be clinically significant);
* Major trauma or major surgery within 3 months prior to screening, or planned surgery during the study;
* Donation or blood loss ≥ 400 mL, or received blood transfusion within 12 weeks prior to screening; Or blood donation or blood loss ≥ 200 mL within 1 month prior to screening;
* Participants who are participating in another clinical trial, or have not undergone a protocol-specified washout period prior to this study;
* Received any antisense oligonucleotides (ASO) or using any small molecule interfering ribonucleic acid (siRNA) drug within 12 months prior to screening;
* Participants with abnormal thyroid function judged by the investigator to be ineligible for enrollment;
* Obviously abnormal laboratory test results;
* History of vasculitis or signs and symptoms of underlying vasculitis;
* Any other circumstance or condition that, in the opinion of the investigator, the participants are inappropriate for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with serum HBsAg < limit of detection (LOD) 0.05 international unit per milliliter (IU/mL) and Hepatitis B Virus (HBV) DNA < lower limit of quantification (LLOQ) with or without HBsAb seroconversion. | Up to 24 weeks

SECONDARY OUTCOMES:
Number and percentage of participants with serum HBsAg < LOD and/or HBV DNA < LLOQ. | Up to 48 weeks
Proportion of participants maintaining sustained response; | Up to 48 weeks
The changes of liver HBsAg, HBcAg, HBV RNA, integration HBV DNA and covalently closed circular DNA (cccDNA) compared to baseline; | Up to 48 weeks
The changes in the phenotype of liver immune cells compared to baseline; | Up to 48 weeks
The changes of peripheral blood cytokines compared to baseline; | Up to 48 weeks
The changes of peripheral blood immune cell phenotypes compared to baseline; | Up to 48 weeks
The changes of serum HBsAg, HBsAb, HBV DNA, HBV RNA, HBeAg, HBeAb compared to baseline; | Up to 48 weeks
The changes in peripheral blood metabolomics compared to baseline; | Up to 48 weeks
The changes in peripheral blood proteomics compared to baseline; | Up to 48 weeks
The changes in liver metabolomics compared to baseline, if applicable ; | Up to 48 weeks
AHB-137 drug concentrations, and metabolite profiling, if applicable; | Up to 48 weeks
Number and percentage of participants with detectable anti-drug antibodies (ADA); | Up to 48 weeks
Safety: Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAE) and clinically significant examination results. | Up to 48 weeks
  Examination including laboratory examination, electrocardiogram (ECG) examination.

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Zhang, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No